CLINICAL TRIAL: NCT01895348
Title: A Comparison of Surgical Outcome Following Drug-induced Sleep Endoscopic Diagnosis Using Propofol or Dexmedetomidine for Sedation : A Prospective Randomized Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2012-0291
Record Dates: First submitted 2013-06-19; First posted 2013-07-10 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- propofol only (Active Comparator)
  Interventions: Drug: Propofol
- propofol-remifentanil (Active Comparator)
  Interventions: Drug: propofol-remifentanil
- dexmedetomidine-remifentanil (Active Comparator)
  Interventions: Drug: Dexmedetomidine-remifentanil

INTERVENTIONS:
Drug: Propofol — Propofol TCI: effect-site concentration(Ce): Ce was titrated to 1.0 μg/ml and increased by 0.2 μg/ml every five minutes
  Arms: propofol only
Drug: propofol-remifentanil — Propofol TCI: effect-site concentration(Ce): Ce was titrated to 1.0 μg/ml and increased by 0.2 μg/ml every five minutes Remifentanil TCI: effect-site concentration(Ce): Ce was titrated to 1.5 μg/ml
  Arms: propofol-remifentanil
Drug: Dexmedetomidine-remifentanil — Dexmedetomidine infusion: After the loading dose (1 mcg/kg for 10 minutes), the continuous infusion was done (0.2 mcg/kg/hr) and the infusion rate was increased by 0.2 mcg/kg/hr every five minutes (maximum infusion rate: 1.4 mcg/kg/hr) Remifentanil TCI: effect-site concentration(Ce): Ce was titrated to 1.5 μg/ml
  Arms: dexmedetomidine-remifentanil

SUMMARY:
Obstructive sleep apnea is a common disease, associated with cardiovascular disease, cerebrovascular disease, and many other medical conditions. Therefore the precise diagnosis and treatment are important. With drug-induced sleep endoscopy (DISE), the three-dimensional evaluation of upper airway and airway obstruction could be possible. The problem of the DISE is that there is the difference between a sedative-induced sleep and normal sleep. Moreover there were no standard sedation protocol of DISE. Propofol has short half-life, about 3 minutes, so the patients could recover quickly from it. In recent years, using target controlled infusion(TCI) of propofol, the effective effect-site concentration for DISE could be reached easily with hemodynamic stability and minimal toxic effect. In a previous pilot study, the endoscopy for the diagnosis of sleep apnea could be done successfully with propofol TCI. However there were some desaturation events, although the EEG showed that the patient was not in deep sleep enough. Therefore we thought that not only further study of propofol for DISE but also the study of other drugs for DISE will be needed to overcome this limitation. Dexmedetomidine, the selective α2-adrenoreceptor agonist, has analgesic effect and almost no respiratory depression, therefore it could be a good alternative drug for DISE. The purpose of this study is designing the appropriate sedation protocol for DISE using propofol or dexmedetomidine, and enabling the safer and more accurate DISE.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1, 2
* Age ≥ 20 yrs
* undergoing drug-induced endoscopy

Exclusion Criteria:

* patient's reject
* patients with hearing impairment or neurological deficits
* patients taking medicine that can affect the central nervous system
* History of adverse drug reactions
* Glasgow coma scale ≤ 15
* could not undergo the endoscopy
* could undergo the endoscopy, but do not undergo UPPP

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Desaturation rate | Baseline / 5 min after remifentanil TCI start / 5 min after propofol TCI start or 10 min after dexmedetomidine loading start / every 5 min until surgeon can do endoscopy successfully / immediately after endoscopy
  SpO2 < 90% (checked by pulse oximetry)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea